CLINICAL TRIAL: NCT04466813
Title: Effects of Dry Needling on Stiffness in Latent Trigger Points a Randomized Controlled Trial
Brief Title: Effect of Dry Needling on Muscle Mechanical Properties and Muscle Contractility in Latent Trigger Points
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Castilla-La Mancha (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DNMYOTMG
Record Dates: First submitted 2020-07-06; First posted 2020-07-10 (Actual); Last update posted 2020-10-23 (Actual); Status verified 2020-07

CONDITIONS: Trigger Point Pain, Myofascial
Keywords: Latent trigger point; Dry needling; Myotonometer; Tensiomyography
MeSH Terms: conditions — Myofascial Pain Syndromes

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Deep Dry Needling (Experimental): Intervention-Dry Needling: Deep Dry Needing into the latent trigger point of the upper trapezius muscle
  Interventions: Device: Intervention-Dry Needling
- Sham Dry Needling (Sham Comparator): Control-Dry Needling: Sham Dry Needling into the latent trigger point of the upper trapezius muscle
  Interventions: Device: Control-Dry Needling

INTERVENTIONS:
Device: Intervention-Dry Needling — Deep Dry Needling into the site of the latent Trigger Point of the upper trapezius muscle.
  1 session in upper trapezius muscle moving the needle up and down ten times.
  Arms: Deep Dry Needling
Device: Control-Dry Needling — Sham Dry Needling into the site of the latent Trigger Point of the upper trapezius muscle with non-penetrating needles
  Arms: Sham Dry Needling

SUMMARY:
The purpose of this study is to determine whether application of Dry Needling (DN) is effective for improved Muscle Mechanical Properties and Muscle Contractility in Latent Trigger Points point (LTrP) of upper trapezius. Randomized controlled trial, in parallel with cross-control design. Two groups with LTrP in upper trapezius, and will be randomly selected to DN group or Sham-Dn group.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 30 years
* The presence of LTrP in the middle third of the upper trapezius muscle on the dominant side
* Being able to provide written informed consent
* Being able to follow instructions and realize clinical tests

Exclusion Criteria:

* Any pharmacological therapeutic
* Any medical treatment or physical therapies at cervical region during the 6-month before this study - Any diagnosed health problem
* Any history of head and upper extremity surgery or trauma
* Any red flags to DN, (ie: metabolic diseases, pregnancy, kinesiophobia, Infection, cancer)
* Absence of recurrent history of neck pain
* No neck pain symptomatology the previous 6 months
* Cervical disk herniation

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2020-07-20 (Actual); Primary Completion 2020-09-20 (Actual); Study Completion 2020-10-20 (Actual)

PRIMARY OUTCOMES:
Change in Stiffness | Baseline, at 30 minutes after treatment, at 24 hours after treatment, at 72 hours after treatment
  This outcome measure is obtained by a device named MyotonPro. Stiffness reflects the resistance of the muscle to the force deforming the muscle.
Change in Maximal Radial Displacement (Dm) | Baseline, at 30 minutes after treatment, at 24 hours after treatment, at 72 hours after treatment
  This outcome measure is obtained by a device named Tensiomiography. The variable Dm is given by the radial displacement of the muscular belly in a transverse plane, expressed in millimeters (mm) and depends on muscle tone or stiffness. A low Dm is related to a high muscle tone or an excess of stiffness, while a high Dm value indicates a lack of muscle tone or stiffness defect.

SECONDARY OUTCOMES:
Change in Oscillation Frequency | Baseline, at 30 minutes after treatment, at 24 hours after treatment, at 72 hours after treatment
  This outcome measure is obtained by a device named MyotonPro. The frequency of the damped oscillations characterizes the muscle tone.
Change in Decrement (elasticity) | Baseline, at 30 minutes after treatment, at 24 hours after treatment, at 72 hours after treatment
  This outcome measure is obtained by a device named MyotonPro.The logarithmic decrement of the damping oscillations characterizes muscle elasticity which is the ability of the muscle to restore its initial shape after contraction
Change in Mechanical Stress Relaxation Time [ms] | Baseline, at 30 minutes after treatment, at 24 hours after treatment, at 72 hours after treatment
  This outcome measure is obtained by a device named MyotonPro. Mechanical Stress Relaxation Time [ms] is the time for a muscle to recover tis shape from deformation after a voluntary contraction or a removal of an external force.
Change in Ratio of deformation and Relaxation time, characterising Creep (Deborah number) | Baseline, at 30 minutes after treatment, at 24 hours after treatment, at 72 hours after treatment
  This outcome measure is obtained by a device named MyotonPro. Ratio of deformation and Relaxation time, characterising Creep (Deborah number) is the gradual elongation of a tissue over time when placed under a constant tensile stress.
Change in Contraction time (Tc) | Baseline, at 30 minutes after treatment, at 24 hours after treatment, at 72 hours after treatment
  This outcome measure is obtained by a device named Tensiomiography. Contraction time (Tc) as a time between 10% and 90% of the contraction
Change in Delay time (Td) | Baseline, at 30 minutes after treatment, at 24 hours after treatment, at 72 hours after treatment
  This outcome measure is obtained by a device named Tensiomiography. Delay time (Td) as a time between the electrical impulse and 10% of the contraction
Change in Sustain time (Ts) | Baseline, at 30 minutes after treatment, at 24 hours after treatment, at 72 hours after treatment
  This outcome measure is obtained by a device named Tensiomiography. Sustain time (Ts) as a time between 50% of the contraction and 50% of the relaxation
Change in Relaxation time (Tr) | Baseline, at 30 minutes after treatment, at 24 hours after treatment, at 72 hours after treatment
  This outcome measure is obtained by a device named Tensiomiography. Relaxation time (Tr) as a time between 90% and 50% of the relaxation
Change in Pressure Pain Perception (PPP) | Baseline, at 30 minutes after treatment, at 24 hours after treatment, at 72 hours after treatment
  Change in Pain Pressure Threshold (PPT) as assessed using an manual mechanical algometer. The procedure performed was the same as the prior described, but pressure was kept until 2.5 kg/cm2 and maintained for 5 seconds, whereas the subject had to characterize the level of pain using a 10-mm visual analog scale (VAS)

CONTACTS AND LOCATIONS:
Overall Officials: Javier Abián-Vicén, PhD, Study Director — Castilla-La Mancha University
Locations (1):
- Performance and Sport Rehabilitation Laboratory, Toledo, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sanchez-Infante J, Bravo-Sanchez A, Jimenez F, Abian-Vicen J. Effects of dry needling on mechanical and contractile properties of the upper trapezius with latent myofascial trigger points: A randomized controlled trial. Musculoskelet Sci Pract. 2021 Dec;56:102456. doi: 10.1016/j.msksp.2021.102456. Epub 2021 Sep 3. PMID 34507046